CLINICAL TRIAL: NCT01405768
Title: A Randomized Trial of Buffered vs Nonbuffered Lidocaine With Epinephrine for Cervical Loop Excision
Brief Title: Buffered Lidocaine for Loop Electrosurgical Excision Procedures (LEEPs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201104269
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-06

CONDITIONS: Uterine Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Arm (Active Comparator): Women in this arm will receive plain lidocaine with epinephrine injected into their cervix prior to the LEEP procedure.
  Interventions: Drug: Non-buffered lidocaine
- Buffered Lidocaine (Experimental): Women in this arm will receive sodium bicarbonate buffered lidocaine mixed with epinephrine injected into their cervix prior to the LEEP procedure.
  Interventions: Drug: sodium bicarbonate buffered lidocaine

INTERVENTIONS:
Drug: sodium bicarbonate buffered lidocaine — 8.4% sodium bicarbonate will be mixed with lidocaine in a 1:10 ratio prior to mixing with epinephrine and injecting into the cervix.
  Arms: Buffered Lidocaine
Drug: Non-buffered lidocaine
  Arms: Lidocaine Arm

SUMMARY:
Women undergoing a LEEP procedure who receive lidocaine buffered with sodium bicarbonate for their cervical block will experience less injection pain than women who receive plain lidocaine.

DETAILED DESCRIPTION:
Specific aims:

1. To determine whether buffering the agent used for intracervical anesthetic at the time of cervical loop excision reduces injection-related pain. (Hypothesis: buffering significantly reduces injection-related pain.)
2. To determine whether other components of pain from LEEP (procedural pain, and cramping) can be reduced by buffering of intracervical anesthetic among women undergoing cervical loop excision. (Hypothesis: only injection pain will be reduced by buffering, as procedural pain will be reduced by lidocaine equally in both arms and cramping will not be reduced in either arm.)

Background:

Although cervical cancer rates have been dramatically reduced by Pap test screening and the eradication of precursors, more than 100,000 U.S. women develop premalignant cervical lesions each year that require treatment (1). The cervical loop electrosurgical excision procedure (LEEP) is the most common therapy for CIN among U.S. gynecologists. LEEP is performed using one or more 1-2 cm electrosurgical diathermy loops to excise involved and at-risk cervical epithelium including underlying stroma containing glands. Destroying this tissue eliminates cells infected with human papillomavirus, the proximate cause of cervical cancer, and radically reduces the risk of later developing cervical cancer (2, 3).

LEEP is usually performed as an outpatient procedure using intracervical anesthesia, most commonly combining lidocaine as an anesthetic agent with epinephrine as a hemostatic agent; final hemostasis is achieved using electrosurgical fulguration and topical hemostatic agents (4). Prior literature has suggested that pain from LEEP has 3 components: pain from injection of the anesthetic combination, pain from the excision, and cramping from reflex uterine contractions (5). While cramping can be controlled with oral nonsteroidal anti-inflammatory agents, injection and procedural pain are not. Most women categorize the pain of LEEP as 3-7 on a 0-10 Likert scale (5, 6).

Studies of dermal and ocular anesthesia and bone marrow biopsy have found that buffering of acidic local anesthetic agents reduces injection pain (7-14), with up to 66% reduction in pain and significant results in randomized trials involving 30-50 participants. However, the use of buffered lidocaine has not yet been tested for LEEPs. The principal investigator has used both forms of anesthesia and considers both acceptable forms of therapy; he is unaware of any evidence to support the superiority of either arm.

ELIGIBILITY:
Inclusion Criteria:

* antecedent biopsy read as

  * cervical intraepithelial neoplasia (CIN) grade 2 or 3 or microinvasive cancer
  * adenocarcinoma in situ
  * persistent CIN 1
* antecedent pap read as

  * high grade squamous intraepithelial lesion
  * atypical glandular cells
  * persistent low grade squamous intraepithelial lesion

Exclusion Criteria:

* anatomy unsuitable for safe office loop excision based on operator judgement
* inability to tolerate procedure under local anesthesia
* pregnancy
* age less than 18 years
* inability to understand spoken or written English
* refusal of consent
* prisoner
* mental incapacity
* anticoagulant or antiplatelet therapy, or known bleeding diathesis
* use of analgesics other than over the counter medications(OTC meds include NSAIDS or Tylenol) within 7 days of scheduled LEEP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Stewart Massad, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Ruegg TA, Curran CR, Lamb T. Use of buffered lidocaine in bone marrow biopsies: a randomized, controlled trial. Oncol Nurs Forum. 2009 Jan;36(1):52-60. doi: 10.1188/09.ONF.52-60. PMID 19136338
- [Background] Sharma T, Gopal L, Shanmugam MP, Bhende P, George J, Samanta TK, Mukesh BN. Comparison of pH-adjusted bupivacaine with a mixture of non-pH-adjusted bupivacaine and lignocaine in primary vitreoretinal surgery. Retina. 2002 Apr;22(2):202-7. doi: 10.1097/00006982-200204000-00011. PMID 11927854
- [Background] Fitton AR, Ragbir M, Milling MA. The use of pH adjusted lignocaine in controlling operative pain in the day surgery unit: a prospective, randomised trial. Br J Plast Surg. 1996 Sep;49(6):404-8. doi: 10.1016/s0007-1226(96)90011-9. PMID 8881789
- [Background] Burns CA, Ferris G, Feng C, Cooper JZ, Brown MD. Decreasing the pain of local anesthesia: a prospective, double-blind comparison of buffered, premixed 1% lidocaine with epinephrine versus 1% lidocaine freshly mixed with epinephrine. J Am Acad Dermatol. 2006 Jan;54(1):128-31. doi: 10.1016/j.jaad.2005.06.043. PMID 16384767
- [Background] Younis I, Bhutiani RP. Taking the 'ouch' out - effect of buffering commercial xylocaine on infiltration and procedure pain - a prospective, randomised, double-blind, controlled trial. Ann R Coll Surg Engl. 2004 May;86(3):213-7. doi: 10.1308/003588404323043382. PMID 15140310
- [Background] Masters JE. Randomised control trial of pH buffered lignocaine with adrenaline in outpatient operations. Br J Plast Surg. 1998 Jul;51(5):385-7. doi: 10.1054/bjps.1997.0293. PMID 9771366
- [Background] Orlinsky M, Hudson C, Chan L, Deslauriers R. Pain comparison of unbuffered versus buffered lidocaine in local wound infiltration. J Emerg Med. 1992 Jul-Aug;10(4):411-5. doi: 10.1016/0736-4679(92)90269-y. PMID 1430977
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine Arm | Buffered Lidocaine
Started | 28 | 28
Completed | 24 | 28
Not Completed | 4 | 0
Not completed — Didn't complete questionnaire correctly | 4 | 0

BASELINE CHARACTERISTICS:
Population: 4 women from the lidocaine arm who did not complete the questionnaire correctly were excluded from analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Arm | Buffered Lidocaine | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.3) | 32.3 (7.6) | 32.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 13 | 12 | 25
  White | 10 | 14 | 24
  Hispanic/Latina | 0 | 1 | 1
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52
Parity [Number; unit: participants] — Parity indicates the number of >20-week births (including viable and non-viable; i.e., stillbirths). Pregnancies consisting of multiples, such as twins or triplets, count as one birth for the purpose of this notation.
  participants
    0 | 3 | 6 | 9
    1 | 5 | 7 | 12
    2+ | 16 | 15 | 31
Indication [Number; unit: participants] — HSIL = High grade squamous intraepithelial lesion
  CIN 2 = Cervical squamous intraepithelial neoplasia 2
  CIN 3 = Cervical squamous intraepithelial neoplasia 2
  AIS = Adenocarcinoma in situ
  Persistent CIN 1 = Persistent cervical squamous intraepithelial neoplasia 1
  participants
    HSIL | 8 | 4 | 12
    CIN 2 | 4 | 7 | 11
    CIN 3 | 11 | 15 | 26
    AIS | 1 | 1 | 2
    Persistent CIN 1 | 0 | 1 | 1
Procedure type [Number; unit: participants]
  Ectocervix only | 16 | 17 | 33
  Ectocervix and endocervix | 8 | 11 | 19
Number of passes [Number; unit: participants]
  1 | 6 | 11 | 17
  2 | 12 | 12 | 24
  3+ | 6 | 5 | 11
Ectocervical loop size (in mm) [Number; unit: participants]
  15 x 12 | 3 | 7 | 10
  20 x 12 | 13 | 16 | 29
  Other | 8 | 5 | 13
Endocervical loop size (in mm) [Number; unit: participants] — 8 patients in the Lidocaine arm had the endocervical loop used.
  11 patients in the Buffered Lidocaine arm had the endocervical loop used.
  participants
    10 x 10 | 5 | 11 | 16
    15 x 12 | 2 | 0 | 2
    10 x 8 | 1 | 0 | 1
Estimated blood loss (in mL) [Number; unit: participants]
  0 mL | 3 | 6 | 9
  1-5 mL | 9 | 8 | 17
  6-10 mL | 7 | 9 | 16
  >10 mL | 5 | 5 | 10
Anesthetic volume (in mL) [Number; unit: participants]
  6-9 mL | 12 | 11 | 23
  10 mL | 11 | 15 | 26
  >10 mL | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Injection Pain Score (Mean)
Description: A Likert visual analog scale will be used to document each study participant's level of pain experienced during injection of the cervical block.
  Within 30 minutes of completion of the procedure and after instruction by the investigators, women reported the intensity of their pain by marking single lines across 100-mm Likert visual analog scales. Scales did not include hashmarks or internal descriptors, as these have been shown to bias responses and diminish reliability.
  Patient marks on 100-mm Likert scale lines were measured, and a score was determined by the length marked off in millimeters. Patients who wrote "no pain" were considered to have marked 0 mm.
Time Frame: Within 30 minutes of completion of procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Arm | Buffered Lidocaine
Number analyzed (Participants) | 24 | 28
units on a scale | 25 (19) | 19 (17)
Statistical Analysis 1: Comparison: Lidocaine Arm vs Buffered Lidocaine; Test type: Superiority or Other; p = .13, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Overall LEEP Procedure Pain Including Procedural Pain and Cramping (Mean)
Description: A Likert visual analog scale will be used to determine the overall pain experienced by each study participant including injection pain, procedural pain, and cramping.
  Within 30 minutes of completion of the procedure and after instruction by the investigators, women reported the intensity of their pain by marking single lines across 100-mm Likert visual analog scales. Scales did not include hashmarks or internal descriptors, as these have been shown to bias responses and diminish reliability.
  Patient marks on 100-mm Likert scale lines were measured, and a score was determined by the length marked off in millimeters. Patients who wrote "no pain" were considered to have marked 0 mm.
Time Frame: Within 30 minutes of completion of procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Arm | Buffered Lidocaine
Number analyzed (Participants) | 24 | 28
units on a scale
  Injection pain | 25 (19) | 19 (17)
  Procedure pain | 27 (18) | 19 (17)
  Cramping pain | 19 (16) | 18 (16)

3. Primary Outcome: Injection Pain Score (Median)
Description: as for outcome 1
Time Frame: Within 30 minutes of completion of the procedure
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lidocaine Arm | Buffered Lidocaine
Number analyzed (Participants) | 24 | 28
units on a scale | 26 [0 to 75] | 18 [0 to 60]
Statistical Analysis 1: Comparison: Lidocaine Arm vs Buffered Lidocaine; Test type: Superiority or Other; p = .13, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Overall LEEP Procedure Pain Including Procedural Pain and Cramping (Median)
Description: as for outcome 2
Time Frame: Within 30 minutes of completion of procedure
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lidocaine Arm | Buffered Lidocaine
Number analyzed (Participants) | 24 | 28
units on a scale
  Injection pain | 26 [0 to 75] | 18 [0 to 60]
  Procedure pain | 25 [0 to 63] | 13 [0 to 54]
  Cramping pain | 19 [0 to 62] | 14 [0 to 65]

ADVERSE EVENTS:
Time Frame: Start of procedures through 30 days after completion of procedure. The procedure occurs on Day 1.
Arm/Group | Lidocaine Arm | Buffered Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

LIMITATIONS AND CAVEATS:
* Small sample - may have missed a significant difference when one really exists
* Procedures performed by 2nd year residents vs. procedure performed by more skilled surgeon (less pain)
* Used needle extenders/27-gauge needles vs. Potocki needles

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes